CLINICAL TRIAL: NCT01263158
Title: Labour Augmentation by Means of Oxytocin - Obstetric Outcome and Women's Experiences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Ryhov County Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: L586-97
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Slow Labour Progress
Keywords: randomised controlled trial; nulliparous women; slow labour progress; prolonged labour; oxytocin augmentation; operative delivery; childbirth experience

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expectant group (Experimental): Arrest in labour progress for 2-3 hours and no progress after amniotomy. Expectancy of standard oxytocin treatment for 3 hours.
  Interventions: Other: Expectancy of standard oxytocin treatment
- Early oxytocin group (No Intervention): Arrest in labour progress for 2-3 hours and no progress after amniotomy. Oxytocin treatment started within 20 minutes.

INTERVENTIONS:
Other: Expectancy of standard oxytocin treatment
  Arms: Expectant group

SUMMARY:
Slow labour progress is common in nulliparous women and is associated with childbirth complications and negative birth experiences. Oxytocin augmentation is widely used to treat slow labour despite associated risks for the fetus. An ongoing debate concerns whether oxytocin should be administered directly or postponed after arrested labour. The overall aim is to study labour progress in healthy nulliparous women and to compare childbirth outcomes and experiences in women randomised to expectant versus early oxytocin augmentation for slow labour progress.

The hypothesis is that it is to early to start oxytocin treatment when labour progress has been slow for 2 to 3 hours in healthy women having their first baby and therefore beneficial for childbirth outcomes to postpone oxytocin for another 3 hours. In this randomised controlled trial nulliparous women with a normal pregnancy, spontaneous onset of active labor at term, and a cervical dilatation of 4 - 9 centimetres on admission to the delivery ward were included (n=2,072). All women whose labour did not progress after amniotomy (n=630) were randomly allocated either to labour augmentation by oxytocin infusion (Early oxytocin, n=314) or to postponement of oxytocin augmentation for another three hours (Expectant, n=316). One month postpartum the women received a postal questionnaire concerning their experiences of labour and birth. All participating women gave their informed consent. Maternal and neonatal outcomes like mode of delivery, postpartum haemorrhage, perinatal lacerations, low Apgar score, need of neonatal intensive care and maternal experiences of childbirth were compared between the randomised groups.

DETAILED DESCRIPTION:
In contemporary handling of labouring women in the western world, it has become extremely common to intervene through "active" or disciplined" management (Enkin et al., Widela et al., Gerdhardstein et al., Frigoletto et al). It is a widespread routine - and potential side effects will therefore have a great impact. The use of the hormone oxytocin to enhance and speed up labour is the most common method, but the sparse scientific data regarding its effect are inconsistent and mostly demonstrate uncertain and sometime side effects (Thornton & Lilford, Frazer 1994, 1998, Cammu & Van Eeckhout).

The effects, when evaluated, are short-term effects of maternal (obstetric) and fetal outcomes. The studies performed have mostly aimed to investigate whether the active management can reduce the rate of caesarean sections. However, in a meta-analysis of four randomised studies of the effects of oxytocin as intervention in spontaneous labour (Frazer), no significant reduction in the incidence of caesarean section, instrumental deliveries, and use of analgetics or hyper stimulation of labour was found. The only statically significant differences were in side effects: an increased incidence of discomfort and of pain in the group given oxytocin. In this meta-analysis, no significant differences in fetal conditions between the groups were found.

Only one of the studies found sought the women's view on the augmentation procedures (Enkin). Over half of the women who were interviewed, said that the oxytocin treatment was unpleasant and indicate that they would like to try without the drug when giving birth the next time. Over 80% felt that it had increased the amount of pain that they had experienced.

In spite of poor evidence of benefits, around half of birth giving women in Sweden receive oxytocin during labour and in some other countries, far more than that (Waldenström, O'Driscoll, Enkin). It has become the standard care of treating labours with slow progress. According to an investigation by the Swedish National Board of Health and Welfare (Socialstyrelsen 1996), the indications for oxytocin use and the amounts administered are not systematically recorded, and the assessments of its effects are even less well recorded. This makes evaluation by using existing documents very unreliable, and randomised controlled studies.

Aims of the study

The aims of the study are:

* To study the effects of oxytocin treatment vs no or delayed oxytocin treatment on the obstetrical and fetal outcome of spontaneous, but prolonged labour. Primary outcome is rate of spontaneous vaginal deliveries. Secondary outcome are length of labour, postpartum haemorrhage, sphincter lacerations, Apgar score, perceived pain and sense of safety.
* To study labour experiences in women exposed to oxytocin treatment vs women without oxytocin treatment.

Methods

The planned study design is a randomised controlled study with healthy women with normal pregnancies and spontaneous labour, where labour progression is deemed to be prolonged.

Inclusion criteria

Healthy women with full-term, normal pregnancies, spontaneous onset of active labour (effaced cervix and minimum 4 cm dilated) and about to give birth to their first child.

Exclusion criteria

Women with multiple pregnancies, complicated pregnancies, maternal disease during pregnancies, ruptured membranes for more than 2 hours before onset of labour contractions, and fetus in breech presentation.

Sample size calculation

A sample size of 247 in each group is needed to show a difference in spontaneous vaginal deliveries from 81,2% to 90% with a 2-sided test, alpha=0,05 and 80% power.

Procedure

Women fulfilling the criteria as described above are regarded as potential study subjects. Information about the study is distributed during the last trimester at the antenatal clinic. On arrival at the delivery ward, all women fulfilling these criteria are again informed about the study and asked for consent to participate. The progression of labour is thoroughly followed and documented for women who have agreed to participate. If the labour is prolonged during the active phase and is classified as inertia, i.e. with no further opening of the cervix for 2 hours or less than 1 cm in 3 hours, the subject are randomly allocated to either labour augmentation by means of oxytocin infusion within twenty minutes (standard care) or to expectancy and observation another 3 hours (experimental group) If the subjects in the experimental group after the 3 hours still do not progress in their labour, a reassessment regarding the need for labour augmentation is done. Women fulfilling inclusion criteria, and who have agreed to participate, but whose labours proceed normally, are followed according the same protocol, hence serving as external controls.

Assessment and follow-up

The handling of the participants will be done according to a standard protocol holding continuous documentation of the progression of labour, of the amount of oxytocin administered, of the analgesia used and of the obstetric outcome (caesarean section, instrumental vaginal delivery, length of labour, Apgar score etc). At the inclusion in the study, the women assess their expectancies, their perceived pain and sense of safety, using a visual analogue scale. Pain and sense of safety is then assessed at several occasions during and after delivery.

In order to study the women's retrospective perceptions of their labour, they receive a questionnaire regarding their perceived experience one month post partum. This instrument focus on perceived pain, perceived safety, perceived participation in decision-making, sense of control and patient satisfaction. This questionnaire also contains questions regarding breast-feeding and a separate part is to be answered by the father. The latter part holding questions about the fathers' levels of preparation for the delivery, and his expectations and experiences as a supportive person in the labour room. A subgroup of the subjects (24 + 24) - oxytocin exposed and unexposed women - will be interviewed at one and four months after birth, using a qualitative interview method.

Assessment of the baby is done at birth through Apgar scoring, fetal pH and base excess from the umbilical cord blood. In addition to this, a subgroup of the neonates will get their motor activity, heart frequency and respiration activity continuously registered during the first night after birth. This is done with the help of a so-called "sleep-box"

Safety

Three hours after the inclusion in the study, a reassessment of the progress of the labour is performed to evaluate whether the progression is satisfactory, or if oxytocin for those assigned to the experimental group is assessed to be required (procedures).

Reassessments are then done regularly with 2-3 hours interval.

Ethics

Making a randomised, clinical study with care/treatment group and non-care/non-treatment group, always raises the question whether it is good ethics or not to abstain from the presently applied care programme. In this case, scientific data regarding the beneficial outcomes are ambiguous and inconsistent, and it is thus not obvious which of the procedures offered is "best" for the woman and the child. With this background, performing the study including well informed subjects and aiming at evaluating effects of standard procedures, must be considered ethically acceptable.

Importance of the study

There are few controlled studies on the effects of the standard procedure of treating slow labour progression with oxytocin and these show conflicting results. Considering this widespread treatment involving large population of women and newborns, it is of great importance to evaluate potential benefits and side effects in controlled studies. Knowledge about this is especially important in the reorganisation and rationing of resources within obstetric services. In the attempts to shorten women's hospital stays, the shortening of duration of labour has sometimes been considered a means to make obstetric care more cost-efficient and this fact makes independent evaluation of the care even more important.

Furthermore, patients have the right to get evidence based care and treatment. This study will hopefully contribute to a better evidence based handling of women in labour who are subjected to secondary inertia, and in addition it will give us more information about fathers' experiences, which will help us enhance the care of the next-to-kin of the labouring woman.

References

Cammu H, Eeckhout E. A randomised controlled study of early versus delayed use of amniotomy and oxytocin infusion in nulliparous labour. Br J Obstet Gynaecol 1996 Apr;103(4):313-8

Elwood JM. Causal relationships in medicine. Oxford medical publications, Oxford University Press, 1992

Enkin M, Keirse MJNC, Chalmers I. A guide to effective care in pregnancy and childbirth. Pp 205-210, 1994, Oxford University Press Fleiss. Statistical methods for rates and proportions. 2nd ED. Wiley, 1981.

Frazer W, Vendittelli F, Krauss I, Breart G. Early augmentation of labour with amniotomy and oxytocin in nulliparous women: a meta-analysis. Br J Obstet Gynaecol 1998Feb;105(2):189-94.

Frazer WD. Early oxytocin to shorten spontaneous labour. In:Keirse MJNC, Renfrew MJ, et al., eds. Pregnancy and childbirth module, Cochrane Databas of Systematic Reviews. (Cochrane updates on disk. The Cochrane Collaboration; Issue 2, Oxford:

Update software, 1995).

Frigoletto FD, Lièberman E, Lang JM, et al. A Clinical trial of active management of labour. NEJM, 1995;333(12):745-50.

Gerhardstein LP, Allswede MT, Sloan CT, et al. Reduction in the rate of cesarean birth with active management of labour and intermediate-dose oxytocin. J Reprod Med 1995;40(1):4-8

Linde A. Active management of labour - positiva och negativa effekter på den normala förlossningen. 10-poängsuppsats, Barnmorskeutbildningen, Vårdhögskolan i Göteborg, Jan 1997

O'Driscoll K, Foley M, Macdonald D. Active management of labour as an alternativ to cesarean section of dystocia. Obstet Gynaecol 1984;63:485-90

SoS-rapport 1996:24 Hur säker är förlossningsvården?

Thornton JG. Active management of labour: current knowledge and research issues. BMJ 1994;309:366-69.

Videla FK, SatinAJ, Barth WH, et al. Trial of labour: A disciplined approach to labour management resulting in a high rate of vaginal delivery. AM J Perinatol 1995 May;12(3):181-4

Waldenström U, Bergman V, Vasell G. The complexity of labour pain: experiences of 278 women. J Psychosom Obstet Gynaecol 1996 Dec;17(4):215-28.

ELIGIBILITY:
Inclusion criteria:

Nulliparity Normal pregnancy 37+0 - 41+6 weeks Single foetus Cephalic presentation Spontaneous onset of active labour Informed consent

Exclusion Criteria:

Prelabour rupture of membranes Serious maternal disease Fetal intrauterine death

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2072 (Actual)
Dates: Start 1998-10; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Mode of delivery (spontaneous vaginal, instrumental vaginal or caesarean delivery)

SECONDARY OUTCOMES:
Postpartum haemorrhage
Sphincter lacerations
Need of neonatal intensive care
Maternal experiences of childbirth

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Health and Care Sciences, University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Result] Dencker A, Berg M, Bergqvist L, Ladfors L, Thorsen LS, Lilja H. Early versus delayed oxytocin augmentation in nulliparous women with prolonged labour--a randomised controlled trial. BJOG. 2009 Mar;116(4):530-6. doi: 10.1111/j.1471-0528.2008.01962.x. PMID 19250364
- [Result] Dencker A, Berg M, Bergqvist L, Lilja H. Identification of latent phase factors associated with active labor duration in low-risk nulliparous women with spontaneous contractions. Acta Obstet Gynecol Scand. 2010 Aug;89(8):1034-9. doi: 10.3109/00016349.2010.499446. PMID 20636242
- [Result] Dencker A, Taft C, Bergqvist L, Lilja H, Berg M. Childbirth experience questionnaire (CEQ): development and evaluation of a multidimensional instrument. BMC Pregnancy Childbirth. 2010 Dec 10;10:81. doi: 10.1186/1471-2393-10-81. PMID 21143961
- [Result] Bergqvist L, Dencker A, Taft C, Lilja H, Ladfors L, Skaring-Thorsen L, Berg M. Women's experiences after early versus postponed oxytocin treatment of slow progress in first childbirth--a randomized controlled trial. Sex Reprod Healthc. 2012 Jun;3(2):61-5. doi: 10.1016/j.srhc.2012.03.003. Epub 2012 Mar 24. PMID 22578752